CLINICAL TRIAL: NCT04216329
Title: A Phase I Clinical Trial of Selinexor (KPT-330) in Combination With Temozolomide and Radiation Therapy in Patients With Newly Diagnosed Glioblastoma
Brief Title: Selinexor (KPT-330) in Combination With Temozolomide and Radiation Therapy in Patients With Newly Diagnosed Glioblastoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kevin Camphausen, M.D., Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 200027; 20-C-0027
Record Dates: First submitted 2019-12-31; First posted 2020-01-02 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Gliosarcoma; Newly Diagnosed; Glioblastoma
Keywords: Radiotherapy; GBM; Gliosarcoma
MeSH Terms: conditions — Gliosarcoma; Glioblastoma | interventions — selinexor; Temozolomide; Serotonin Antagonists; Olanzapine; Salts; Sodium Chloride; Loperamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1/Experimental Therapy - Selinexor with Temozolomide and Radiation (Experimental): Selinexor with temozolomide and radiation
  Interventions: Drug: Selinexor; Drug: Temozolomide; Radiation: Generic Radiation therapy (RT); Other: Selective serotonin receptor (5-HT3) antagonists; Other: Olanzapine; Dietary Supplement: Salt tablets; Other: Anti-diarrheal

INTERVENTIONS:
Drug: Selinexor — Selinexor will be administered orally at an initial dose of 80 mg. The first dose will be given on day 2 of radiation and will thereafter be administered weekly on the second day of weekly radiation on weeks 1, 2, 4, and 5. If this dose level is tolerated, the dose will be escalated to 60 mg twice a week (days 1 and 4) on weeks 1,2,4,5. The third and final dose level will also be 60mg administered twice weekly for 6 weeks starting on days 1 and 4 radiation.
  Other Names: Xpovio
Drug: Temozolomide — Temozolomide will begin on the first day or evening prior of radiation and be administered orally daily at a dose of 75 mg/m^2 during the radiation treatment. Temozolomide will continue until the completion of radiation and then will be stopped. Beginning 1-month post-radiation therapy (RT), the adjuvant temozolomide will be given per standard of care.
  Other Names: Temodar
Radiation: Generic Radiation therapy (RT) — Radiation therapy (RT) will be administered daily (Monday to Friday)
Other: Selective serotonin receptor (5-HT3) antagonists — Anti-emetic for breakthrough nausea.
  Other Names: Serotonin antagonists
Other: Olanzapine — 2.5mg to 5mg once a day if weight loss is rapid.
  Other Names: Zyprexa Relprevv; Zyprexa Zydis; Zyprexa
Dietary Supplement: Salt tablets — To treat hyponatremia, add salt tablets to participants diet per institutional guidelines.
  Other Names: Sodium Chloride tablets
Other: Anti-diarrheal — Treat diarrhea with an anti-diarrheal per institutional guidelines
  Other Names: Loperamide; Imodium

SUMMARY:
Background:

Glioblastoma is a type of brain cancer. Treatments include radiation, chemotherapy, and surgery. But survival rates are poor. Researchers think that the drug selinexor, when combined with chemotherapy and radiation, might help.

Objective:

To learn the highest dose of selinexor that people with brain cancer can tolerate when given with temozolomide and radiation therapy.

Eligibility:

People ages 18 and older with brain cancer that has not been treated with chemotherapy or radiation.

Design:

Participants will be screened under another protocol.

Before participants start treatment, they will have tests:

Neurological and physical evaluations

Blood and urine tests

Possible computed tomography (CT) scan or magnetic resonance imaging (MRI) of the brain if they have not had one in 3 weeks. Participants will lie in a machine that takes pictures of the body. They may have a dye injected into a vein.

Surveys about their well-being

Participants will have radiation to the brain for up to 6 weeks. This will usually be given once a day, Monday through Friday.

Starting the second day of radiation, participants will take selinexor by mouth once a week. They will take it in weeks 1, 2, 4, and 5. The timing may be changed.

Starting the first day of radiation, participants will take temozolomide by mouth once a day until they complete radiation.

Participants will have blood tests once per week during treatment.

Participants will have a follow-up visit 1 month after they complete treatment. Then they will have visits at least every 2 months for the first 2 years, then at least every 3 months for another year. Visits will include MRIs and blood tests.

DETAILED DESCRIPTION:
Background:

* Although radiation has been shown to improve outcomes in patients with glioblastoma (GBM), median survival remains poor. Even with the addition of temozolomide (TMZ) to surgical resection and radiotherapy, most GBMs will recur in field or adjacent to the high dose radiation volume.
* High rates of local failure indicate that GBM cells in situ are relatively radioresistant and that the effectiveness of GBM radiotherapy would benefit from additional radiosensitization.
* Selinexor has recently been shown to enhance the radiosensitivity of glioma cells both in vitro and in vivo.

Objectives:

-Assess the safety, tolerability, and maximum tolerated dose of selinexor when combined with temozolomide and radiotherapy in patients with newly diagnosed glioblastoma and gliosarcoma.

Eligibility:

* Men and women greater than 18 years old
* Histologically confirmed newly diagnosed glioblastoma or gliosarcoma
* Karnofsky Performance Scale (KPS) greater than or equal to 70
* Patients who have not previously been treated with chemotherapy or radiation therapy

Design:

* This is a Phase I trial to determine the safety and tolerability of selinexor in combination with external beam radiation therapy (RT) and temozolomide in patients with newly diagnosed glioblastoma or gliosarcoma using a "3 plus 3 design" and three dose escalation levels, with 3 patients per dose level (provided no dose limiting toxicity (DLT), a maximum of 21 patients will be enrolled.
* Patients will be treated with external beam radiation therapy in a standard manner with temozolomide given daily during radiation. Selinexor will be administered concurrent with the RT/temozolomide.
* We anticipate accrual of 21 evaluable patients which will take approximately 2 years. The accrual ceiling has been set to 24 patients.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Histological diagnosis

     * Pathologically confirmed glioblastoma or gliosarcoma (including astrocytoma, grade IV)
  2. Patients must be eligible for definitive external beam radiotherapy and temozolomide.
  3. Age >18 years. Because no dosing or adverse event data are currently available on the use of Selinexor in combination with Temodar in patients <18 years of age, children are excluded from this study.
  4. Patients should have a Karnofsky performance scale (KPS) greater than or equal to 70
  5. Absolute neutrophil count (ANC) >1.5x10^9/L; platelet count >100x10^9/L; and hemoglobin (Hb) >9.0 g/dL. Note: the use of transfusion or other intervention prior to cycle 1 day 1 to achieve Hb >9.0 g/dL is acceptable.
  6. Ability of subject or Legally Authorized Representative (LAR) to understand and the willingness to sign a written informed consent document.
  7. The effects of Selinexor on the developing human fetus are unknown. For this reason and because Selinexor agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study treatment and for one month after treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
  8. Patients must have had surgery and/or biopsy not greater than 8 weeks prior to initial evaluation to be eligible for this study.

     EXCLUSION CRITERIA:

  <!-- -->

  1. Patients who are receiving any other investigational agents and have had prior therapy including:

     * Patients who have previously received radiation therapy (RT) to the brain.
     * Patients who received chemotherapy for the treatment of their glioma
     * Patients who are being treated with implanted Gliadel wafers
     * Patients who are being treated with tumor treating fields.
  2. History of allergic reactions attributed to compounds of similar chemical or biologic composition to selinexor or temozolomide used in study.

  3 Patients with coagulation problems and medically significant bleeding in the month prior to start of treatment (peptic ulcers, epistaxis, spontaneous bleeding). Prior history of deep vein thrombosis (DVT) or pulmonary embolism (PE) is not exclusionary.

  4. Patients with active uncontrolled or suspected infections

  5. Patients with severe liver dysfunction defined as:
  * Total bilirubin > 1.5 x upper limit of normal (ULN) Note: Subjects with Gilberts syndrome should not be excluded as long as total bilirubin is < 3.0 x ULN and documentation to support diagnosis is available.
  * Serum glutamate pyruvate transaminase (SGPT) or called as Alanine aminotransferase (ALT) greater than or equal to 3 x ULN = 135 U/L; for the purpose of this study, the ULN for SGPT is 45 U/L
  * Serum glutamic oxaloacetic transaminase (SGOT) or called as Aspartate aminotransferase (AST) greater than or equal to 3 x ULN = 150 U/L; for the purpose of this study, the ULN for SGOT is 50 U/L
  * Serum albumin greater than or equal to 2 x ULN

    6. Known active hepatitis A, B, or C infection

    7. Human immunodeficiency virus (HIV) patients are not eligible because of their immunocompromised status and overlap of side effects between highly active antiretroviral therapy (HAART) and radiation therapy.

    8 Patients must not have significantly diseased or obstructed gastrointestinal tract malabsorption, uncontrolled vomiting or diarrhea, or inability to swallow oral medication.

    9. Pregnant women are excluded from this study because Selinexor could have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Selinexor, breastfeeding should be discontinued if the mother is treated with Selinexor. These potential risks may also apply to temozolomide used in this study.

    10. Patients with pre-existing known or suspected radiation sensitivity syndromes will be excluded due to potential confounding effect on outcome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2028-07-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin A Camphausen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. All collected IPD will be shared with collaborators under the terms of collaborative agreements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-C-0027.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were enrolled in Dose Level -1.
Groups:
- Dose Level -1: Selinexor 80mg on Weeks 1, 4 With Temozolomide & Radiation: Participants with newly diagnosed glioblastoma or gliosarcoma.
  Selinexor with temozolomide and radiation. Dose Level -1: Selinexor 80mg on Weeks 1, 4
  Temozolomide will begin on the first day or evening prior of radiation and be administered orally daily at a dose of 75 mg/m^2 during the radiation treatment. Temozolomide will continue until the completion of radiation and then will be stopped. Beginning 1-month post-radiation therapy (RT), the adjuvant temozolomide will be given per standard of care.
- Dose Level 1: Selinexor 80mg on Weeks 1, 2, 4, 5 With Temozolomide & Radiation: Participants with newly diagnosed glioblastoma or gliosarcoma.
  Selinexor with temozolomide and radiation. Dose Level 1: Selinexor 80mg on Weeks 1, 2, 4, 5
  Temozolomide will begin on the first day or evening prior of radiation and be administered orally daily at a dose of 75 mg/m^2 during the radiation treatment. Temozolomide will continue until the completion of radiation and then will be stopped. Beginning 1-month post-radiation therapy (RT), the adjuvant temozolomide will be given per standard of care.
- Dose Level 2: Selinexor 60mg Twice a Week on Weeks 1, 2, 4, 5 With Temozolomide & Radiation: Participants with newly diagnosed glioblastoma or gliosarcoma.
  Selinexor with temozolomide and radiation. Dose Level 2: 60mg Twice a Week on Weeks 1, 2, 4, 5
  Temozolomide will begin on the first day or evening prior of radiation and be administered orally daily at a dose of 75 mg/m^2 during the radiation treatment. Temozolomide will continue until the completion of radiation and then will be stopped. Beginning 1-month post-radiation therapy (RT), the adjuvant temozolomide will be given per standard of care.
- Dose Level 3: Selinexor 60mg Twice a Week, Weeks 1-6 With Temozolomide & Radiation: Participants with newly diagnosed glioblastoma or gliosarcoma.
  Selinexor with temozolomide and radiation. Dose Level 3: 60mg Twice a Week, Weeks 1-6
  Temozolomide will begin on the first day or evening prior of radiation and be administered orally daily at a dose of 75 mg/m^2 during the radiation treatment. Temozolomide will continue until the completion of radiation and then will be stopped. Beginning 1-month post-radiation therapy (RT), the adjuvant temozolomide will be given per standard of care.
Period: Overall Study
Arm/Group | Dose Level -1: Selinexor 80mg on Weeks 1, 4 With Temozolomide & Radiation | Dose Level 1: Selinexor 80mg on Weeks 1, 2, 4, 5 With Temozolomide & Radiation | Dose Level 2: Selinexor 60mg Twice a Week on Weeks 1, 2, 4, 5 With Temozolomide & Radiation | Dose Level 3: Selinexor 60mg Twice a Week, Weeks 1-6 With Temozolomide & Radiation
Started | 0 | 3 | 6 | 2
Completed | 0 | 3 | 6 | 2
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants were enrolled in Dose Level -1.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level -1: Selinexor 80mg on Weeks 1, 4 With Temozolomide & Radiation | Dose Level 1: Selinexor 80mg on Weeks 1, 2, 4, 5 With Temozolomide & Radiation | Dose Level 2: Selinexor 60mg Twice a Week on Weeks 1, 2, 4, 5 With Temozolomide & Radiation | Dose Level 3: Selinexor 60mg Twice a Week, Weeks 1-6 With Temozolomide & Radiation | Total
Number analyzed (Participants) | 0 | 3 | 6 | 2 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0 | 0 | 0
  Between 18 and 65 years |  | 3 | 5 | 2 | 10
  >=65 years |  | 0 | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 54.33 (9.29) | 61 (5.66) | 57 (5.66) | 58.45 (6.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 3 | 3 | 1 | 7
  Male |  | 0 | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 0 | 0 | 0 | 0
  Not Hispanic or Latino |  | 3 | 6 | 2 | 11
  Unknown or Not Reported |  | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0 | 0 | 0
  Asian |  | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0 | 0 | 0
  Black or African American |  | 0 | 0 | 0 | 0
  White |  | 3 | 6 | 2 | 11
  More than one race |  | 0 | 0 | 0 | 0
  Unknown or Not Reported |  | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 3 | 6 | 2 | 11

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Selinexor
Description: The MTD is the dose level at which no more than 1 of up to 6 participants experience dose limiting-toxicity (DLT) within 1 month of completion of treatment, and the dose below that at which at least 2 (of< =6) participants have DLT as a result of selinexor/radiation therapy (RT)/temozolomide.
Time Frame: 7 weeks
Measure: Number; unit: mg/m^2
Groups:
- All Participants: All participants who received Selinexor with temozolomide and radiation.
  Selinexor: Selinexor will be administered orally at an initial dose of 80 mg. The first dose will be given on day 2 of radiation and will thereafter be administered weekly on the second day of weekly radiation on weeks 1, 2, 4, and 5. If this dose level is tolerated, the dose will be escalated to 60 mg twice a week (days 1 and 4) on weeks 1,2,4,5. The third and final dose level will also be 60mg administered twice weekly for 6 weeks starting on days 1 and 4 radiation.
  Temozolomide: Temozolomide will begin on the first day or evening prior of radiation and be administered orally daily at a dose of 75 mg/m^2 during the radiation treatment. Temozolomide will continue until the completion of radiation and then will be stopped. Beginning 1-month post-radiation therapy (RT), the adjuvant temozolomide will be given per standard of care.
  Generic Radiation therapy (RT): Radiation therapy (RT) will be administered daily (Monday to Friday)
  Selective serotonin receptor (5-HT3) antagonists: Anti-emetic for breakthrough nausea.
  Olanzapine: 2.5mg to 5mg once a day if weight loss is rapid.
  Salt tablets: To treat hyponatremia, add salt tablets to participants diet per institutional guidelines.
  Anti-diarrheal: Treat diarrhea with an anti-diarrheal per institutional guidelines
Arm/Group | All Participants
Number analyzed (Participants) | 11
mg/m^2 | 60

2. Secondary Outcome: Dose-limiting Toxicities of Selinexor to Concurrent Radiation Therapy and Temozolomide Assessed by the Common Terminology Criteria for Adverse Events (CTCAE) and Radiation Therapy Oncology Group (RTOG)
Description: Dose-limiting toxicities of Selinexor to concurrent radiation therapy and temozolomide. A DLT is defined as a clinically significant adverse event assessed as unrelated to tumor progression, intercurrent illness or concomitant medications and meets any of the criteria such as any Grade 3 or 4 toxicity per Common Terminology Criteria for Adverse Events (CTCAE) v5.0; and any Grade 3 or 4 toxicity per Radiation Therapy Oncology Group (RTOG) acute morbidity. CTCAE: Grade 3 is severe, and Grade 4 is life-threatening. RTOG: Grade 3 Brain/Central nervous system (CNS): neurologic findings present sufficient to require home care; Skin: confluent moist desquamation other than skin folds; Eye: severe keratitis; Ear: severe external otitis; and Grade 4 Brain/CNS is serious neurologic impairment; Skin: ulceration; Eye: loss of vision; and Ear: deafness.DLT's include all adverse events, including clinically significant abnormal findings on laboratory evaluations, regardless of severity.
Time Frame: Measured each week of treatment and up to 30 days post treatment; approximately 6-7 weeks with another month added on = ~ 11 weeks to monitor.
Measure: Number; unit: toxicities
Arm/Group | Dose Level 1: Selinexor 80mg on Weeks 1, 2, 4, 5 With Temozolomide & Radiation | Dose Level 2: Selinexor 60mg Twice a Week on Weeks 1, 2, 4, 5 With Temozolomide & Radiation | Dose Level 3: Selinexor 60mg Twice a Week, Weeks 1-6 With Temozolomide & Radiation
Number analyzed (Participants) | 3 | 6 | 2
toxicities
  Grade 3 DLT - CTCAE | 8 | 19 | 6
  Grade 3 DLT - RTOG | 0 | 0 | 0
  Grade 4 DLT - CTCAE | 1 | 0 | 2
  Grade 4 DLT - RTOG | 0 | 0 | 0

3. Secondary Outcome: Dose-limiting Toxicities Effects on Quality of Life (QOL)
Description: Define the dose-limiting toxicities (DLT) effects on quality of life (QOL) in the setting of the addition of Selinexor to concurrent radiation therapy and temozolomide. A DLT is defined as a clinically significant adverse event assessed as unrelated to tumor progression, intercurrent illness or concomitant medications and meets any of the criteria such as any Grade 3 or 4 toxicity per Common Terminology Criteria for Adverse Events (CTCAE) v5.0; and any Grade 3 or 4 toxicity per Radiation Therapy Oncology Group (RTOG) acute morbidity. QOL life scores will be summarized. DLT's include all adverse events (AE), including clinically significant abnormal findings on laboratory evaluations, regardless of severity. Evaluations completed on participants weekly or complications requiring admission to the emergency room (ER)/hospital are also included in the collection of AEs to determine if DLT.
Time Frame: as for outcome 2
Measure: Number; unit: toxicities
Arm/Group | Dose Level 1: Selinexor 80mg on Weeks 1, 2, 4, 5 With Temozolomide & Radiation | Dose Level 2: Selinexor 60mg Twice a Week on Weeks 1, 2, 4, 5 With Temozolomide & Radiation | Dose Level 3: Selinexor 60mg Twice a Week, Weeks 1-6 With Temozolomide & Radiation
Number analyzed (Participants) | 3 | 6 | 2
toxicities
  Grade 3 DLT-CTCAE | 0 | 0 | 0
  Grade 3 DLT-RTOG | 0 | 0 | 0
  Grade 4 DLT-CTCAE | 0 | 0 | 0
  Grade 4 DLT-RTOG | 0 | 0 | 0

4. Secondary Outcome: Dose-limiting Toxicities (DLT) Effects on Neurocognition
Description: Define the dose-limiting toxicities effects on neurocognition in the setting of the addition of Selinexor to concurrent radiation therapy and temozolomide. A DLT is defined as a clinically significant adverse event assessed as unrelated to tumor progression, intercurrent illness or concomitant medications and meets any of the criteria such as any Grade 3 or 4 toxicity per Common Terminology Criteria for Adverse Events (CTCAE) v5.0; and any Grade 3 or 4 toxicity per Radiation Therapy Oncology Group (RTOG) acute morbidity. DLT's include all adverse events (AE), including clinically significant abnormal findings on laboratory evaluations, regardless of severity. Evaluations completed on participants weekly or complications requiring admission to the emergency room (ER)/hospital are also included in the collection of AE's to determine if DLT.
Time Frame: as for outcome 2
Measure: Number; unit: toxicities
Arm/Group | Dose Level 1: Selinexor 80mg on Weeks 1, 2, 4, 5 With Temozolomide & Radiation | Dose Level 2: Selinexor 60mg Twice a Week on Weeks 1, 2, 4, 5 With Temozolomide & Radiation | Dose Level 3: Selinexor 60mg Twice a Week, Weeks 1-6 With Temozolomide & Radiation
Number analyzed (Participants) | 3 | 6 | 2
toxicities
  Grade 3 DLT-CTCAE | 0 | 0 | 0
  Grade 3 DLT-RTOG | 0 | 00 | 0
  Grade 4 DLT-CTCAE | 0 | 0 | 0
  Grade 4 DLT-RTOG | 0 | 0 | 0

5. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Depression Scale
Description: The PROMIS depression questionnaire in the setting of the addition of Selinexor to concurrent radiation therapy and temozolomide. A DLT is defined as a clinically significant adverse event assessed as unrelated to tumor progression, intercurrent illness or concomitant medications and meets any of the criteria such as any Grade 3 or 4 toxicity per Common Terminology Criteria for Adverse Events (CTCAE) v5.0; and any Grade 3 or 4 toxicity per Radiation Therapy Oncology Group (RTOG) acute morbidity. QOL life scores from questionnaires rating symptoms on a scale of 1 (never) - 5 (very often several times a day) will be summarized. A score of 1 is the best outcome. A score of 5 is worst outcome. The difference between two timepoints - baseline and close of treatment is also reported.
Time Frame: Baseline and completion of treatment, up to 3 years
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | Dose Level 1: Selinexor 80mg on Weeks 1, 2, 4, 5 With Temozolomide & Radiation | Dose Level 2: Selinexor 60mg Twice a Week on Weeks 1, 2, 4, 5 With Temozolomide & Radiation | Dose Level 3: Selinexor 60mg Twice a Week, Weeks 1-6 With Temozolomide & Radiation
Number analyzed (Participants) | 3 | 6 | 2
Score on a scale
  Baseline | 1.63 [1 to 3] | 1.71 [1.125 to 2.625] | 1.71 [1.125 to 2.625]
  Completion of treatment | 1.22 [1 to 1.75] | 2.42 [1 to 3.25] | 2.42 [1 to 3.25]
  Difference between two timepoints | -0.41 [-0.625 to 0.25] | 0.71 [-0.125 to 1.625] | 0.71 [-0.125 to 1.625]
Statistical Analysis 1: Comparison: Dose Level 1: Selinexor 80mg on Weeks 1, 2, 4, 5 With Temozolomide & Radiation; Test type: Other; p = 0.02, Students t-test
Statistical Analysis 2: Comparison: Dose Level 1: Selinexor 80mg on Weeks 1, 2, 4, 5 With Temozolomide & Radiation; Test type: Other; p = 0.07, Students t-test — P-value 0.07 represents the difference between baseline depression scores and completion of treatment scores
Statistical Analysis 3: Comparison: Dose Level 2: Selinexor 60mg Twice a Week on Weeks 1, 2, 4, 5 With Temozolomide & Radiation; Test type: Other; p = 0.02, Students t-test
Statistical Analysis 4: Comparison: Dose Level 2: Selinexor 60mg Twice a Week on Weeks 1, 2, 4, 5 With Temozolomide & Radiation; Test type: Other; p = 0.07, Students t-test — P-value 0.07 represents the difference between baseline depression scores and completion of treatment scores
Statistical Analysis 5: Comparison: Dose Level 3: Selinexor 60mg Twice a Week, Weeks 1-6 With Temozolomide & Radiation; Test type: Other; p = 0.02, Students t-test
Statistical Analysis 6: Comparison: Dose Level 3: Selinexor 60mg Twice a Week, Weeks 1-6 With Temozolomide & Radiation; Test type: Other; p = 0.07, Students t-test — P-value 0.07 represents the difference between baseline depression scores and completion of treatment scores

6. Other Pre Specified Outcome: Dose-limiting Toxicities (DLT) Effects on Quality of Life (QOL) Using the MD Anderson Symptom Inventory for Brain Tumors (MDSAI-BT)
Description: DLT effects on quality of life (QOL) using the MD Anderson Symptom Inventory for Brain Tumors (MDASI-BT) in the setting of the addition of Selinexor to concurrent radiation therapy and temozolomide. A DLT is defined as a clinically significant adverse event assessed as unrelated to tumor progression, intercurrent illness or concomitant medications and meets any of the criteria such as any Grade 3 or 4 toxicity per Common Terminology Criteria for Adverse Events (CTCAE) v5.0; and any Grade 3 or 4 toxicity per Radiation Therapy Oncology Group (RTOG) acute morbidity. QOL life scores from questionnaires rating symptoms on a scale of 0 (symptoms not present)-10 (as bad as you can imagine) will be summarized. A score of 0 is the best outcome. A score of 10 is the worst outcome. The difference between two timepoints - baseline and close of treatment is also reported.
Time Frame: Baseline and close of treatment, up to 3 years
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Dose Level 1: Selinexor 80mg on Weeks 1, 2, 4, 5 With Temozolomide & Radiation | Dose Level 2: Selinexor 60mg Twice a Week on Weeks 1, 2, 4, 5 With Temozolomide & Radiation | Dose Level 3: Selinexor 60mg Twice a Week, Weeks 1-6 With Temozolomide & Radiation
Number analyzed (Participants) | 3 | 6 | 2
Scores on a scale
  Baseline (BL) | 1.21 [0 to 5] | 1.17 [0.678 to 1.857] | 1.17 [0.678 to 1.857]
  Completion of treatment (COT) | 1.6 [0.179 to 3.214] | 1.77 [0.687 to 2.6] | 1.77 [0.687 to 2.6]
  Difference between two timepoints (BL & COT) | 0.39 [0.179 to 1.5] | 0.61 [.006 to 1.072] | 0.61 [.009 to 1.072]

7. Other Pre Specified Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety Scale
Description: The PROMIS anxiety scale in the setting of the addition of Selinexor to concurrent radiation therapy and temozolomide. A DLT is defined as a clinically significant adverse event assessed as unrelated to tumor progression, intercurrent illness or concomitant medications and meets any of the criteria such as any Grade 3 or 4 toxicity per Common Terminology Criteria for Adverse Events (CTCAE) v5.0; and any Grade 3 or 4 toxicity per Radiation Therapy Oncology Group (RTOG) acute morbidity. QOL life scores from questionnaires rating symptoms on a scale of 1 (never) - 5 (always) will be summarized. A score of 1 is the best outcome. A score of 5 is the worst outcome. The difference between two timepoints - baseline and close of treatment is also reported.
Time Frame: Baseline and completion of treatment, up to 3 years
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | Dose Level 1: Selinexor 80mg on Weeks 1, 2, 4, 5 With Temozolomide & Radiation | Dose Level 2: Selinexor 60mg Twice a Week on Weeks 1, 2, 4, 5 With Temozolomide & Radiation | Dose Level 3: Selinexor 60mg Twice a Week, Weeks 1-6 With Temozolomide & Radiation
Number analyzed (Participants) | 3 | 6 | 2
Score on a scale
  Baseline (BL) | 1.63 [1 to 3] | 1.71 [1.125 to 2.625] | 1.71 [1.125 to 2.625]
  Completion of treatment (COT) | 1.22 [1 to 1.75] | 2.42 [1 to 3.25] | 2.42 [1 to 3.25]
  Difference between two timepoints (BL & COT) | -0.41 [-0.625 to 0.25] | 0.71 [-0.125 to 1.625] | 0.71 [-0.125 to 1.625]
Statistical Analysis 1: Comparison: Dose Level 1: Selinexor 80mg on Weeks 1, 2, 4, 5 With Temozolomide & Radiation; Test type: Other; p = 0.09, Students t-test
Statistical Analysis 2: Comparison: Dose Level 2: Selinexor 60mg Twice a Week on Weeks 1, 2, 4, 5 With Temozolomide & Radiation; Test type: Other; p = 0.09, Students t-test
Statistical Analysis 3: Comparison: Dose Level 3: Selinexor 60mg Twice a Week, Weeks 1-6 With Temozolomide & Radiation; Test type: Other; p = 0.09, Students t-test

8. Other Pre Specified Outcome: National Cancer Institute (NCI) Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE)
Description: The NCI PRO-CTCAE in the setting of the addition of Selinexor to concurrent radiation therapy and temozolomide. A DLT is defined as a clinically significant adverse event assessed as unrelated to tumor progression, intercurrent illness or concomitant medications and meets any of the criteria such as any Grade 3 or 4 toxicity per Common Terminology Criteria for Adverse Events (CTCAE) v5.0; and any Grade 3 or 4 toxicity per Radiation Therapy Oncology Group (RTOG) acute morbidity. QOL life scores from questionnaires rating symptoms on a scale of 0 (None) - 4 (Very severe) will be summarized. A score of 0 is the best outcome. A score of 4 is the worst outcome. The difference between two timepoints - baseline and close of treatment is also reported.
Time Frame: Baseline and completion of treatment, up to 3 years
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Dose Level 1: Selinexor 80mg on Weeks 1, 2, 4, 5 With Temozolomide & Radiation | Dose Level 2: Selinexor 60mg Twice a Week on Weeks 1, 2, 4, 5 With Temozolomide & Radiation | Dose Level 3: Selinexor 60mg Twice a Week, Weeks 1-6 With Temozolomide & Radiation
Number analyzed (Participants) | 3 | 6 | 2
Scores on a scale
  Baseline (BL) | 0.29 [0 to 0.85] | 0.53 [0.25 to 0.95] | 0.53 [0.25 to 0.95]
  Completion of treatment (COT) | 0.87 [0.3 to 1.25] | 0.83 [0.684 to 1.05] | 0.83 [0.684 to 1.05]
  Difference between two timepoints (BL & COT) | 0.58 [-0.05 to 1.145] | 0.3 [0.1 to 0.434] | 0.3 [0.1 to 0.434]

9. Other Pre Specified Outcome: Neuro-quality of Life (QOL) Assessment Cognition Function
Description: The Neuro-QOL assessment Cognition Function in the setting of the addition of Selinexor to concurrent radiation therapy and temozolomide. A DLT is defined as a clinically significant adverse event assessed as unrelated to tumor progression, intercurrent illness or concomitant medications and meets any of the criteria such as any Grade 3 or 4 toxicity per Common Terminology Criteria for Adverse Events (CTCAE) v5.0; and any Grade 3 or 4 toxicity per Radiation Therapy Oncology Group (RTOG) acute morbidity. QOL life scores from questionnaires rating symptoms on a scale of 5 (Never) -1 (Very often-several times a day), e.g., thinking slow, will be summarized. A score of 5 is the best outcome. A score of 1 is the worst outcome. The difference between two timepoints - baseline and close of treatment is also reported.
Time Frame: Baseline and completion of treatment, up to 3 years
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | Dose Level 1: Selinexor 80mg on Weeks 1, 2, 4, 5 With Temozolomide & Radiation | Dose Level 2: Selinexor 60mg Twice a Week on Weeks 1, 2, 4, 5 With Temozolomide & Radiation | Dose Level 3: Selinexor 60mg Twice a Week, Weeks 1-6 With Temozolomide & Radiation
Number analyzed (Participants) | 3 | 6 | 2
Score on a scale
  Baseline (BL) | 4.42 [3.125 to 5] | 4.17 [3.625 to 4.5] | 4.17 [3.625 to 4.5]
  Completion of treatment (COT) | 4.39 [2.25 to 5] | 3.67 [3.125 to 4.265] | 3.67 [3.125 to 4.265]
  Difference between two timepoints (BL & COT) | -0.03 [-0.875 to 0.625] | -0.875 [-0.11 to -0.875] | -0.875 [-0.11 to -0.875]

10. Other Pre Specified Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from initiation of treatment on protocol to progression as per Response Assessment in Neuro-Oncology (RANO) criteria or death due to disease progression. Progressive disease is at least two sequential scans separated by at ≥4 weeks both exhibiting ≥25% increase in sum of products of perpendicular diameters or ≥40% increase in total volume of enhancing lesions. Clear clinical deterioration not attributable to other causes apart from tumor or attributable to changes in steroid use. Failure to return for evaluation as a result of death or deteriorating condition.
Time Frame: From initiation of treatment on protocol to progression as per RANO criteria or death due to disease progression, approximately months
Reporting Status: Not Posted, anticipated posting 2028-07

11. Other Pre Specified Outcome: Overall Survival (OS)
Description: OS is defined as the time from initiation of treatment on protocol to date of death due to any cause. For participants alive as of last follow-up, time to death will be censored at last contact date.
Time Frame: From initiation of treatment on protocol to date of death due to any cause, approximately months.
Reporting Status: Not Posted, anticipated posting 2028-07

12. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-Serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned. All adverse events, including clinically significant abnormal findings on laboratory evaluations, regardless of severity, will be followed until return to baseline or stabilization of event.
Time Frame: Adverse events are documented from the first study intervention, Study Day 1, through 30 days after the subject received the last study drug administration, an average of 2.5 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: Selinexor 80mg on Weeks 1, 2, 4, 5 With Temozolomide & Radiation | Dose Level 2: Selinexor 60mg Twice a Week on Weeks 1, 2, 4, 5 With Temozolomide & Radiation | Dose Level 3: Selinexor 60mg Twice a Week, Weeks 1-6 With Temozolomide & Radiation
Number analyzed (Participants) | 3 | 6 | 2
Participants | 3 | 6 | 2

ADVERSE EVENTS:
Time Frame: Adverse events are documented from the first study intervention, Study Day 1, through 30 days after the subject received the last study drug administration, an average of 2.5 months.
Arm/Group | Dose Level 1: Selinexor 80mg on Weeks 1, 2, 4, 5 With Temozolomide & Radiation | Dose Level 2: Selinexor 60mg Twice a Week on Weeks 1, 2, 4, 5 With Temozolomide & Radiation | Dose Level 3: Selinexor 60mg Twice a Week, Weeks 1-6 With Temozolomide & Radiation
All-Cause Mortality (participants affected / at risk) | 1/3 | 5/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/6 | 0/2
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1: Selinexor 80mg on Weeks 1, 2, 4, 5 With Temozolomide & Radiation (N=3) | Dose Level 2: Selinexor 60mg Twice a Week on Weeks 1, 2, 4, 5 With Temozolomide & Radiation (N=6) | Dose Level 3: Selinexor 60mg Twice a Week, Weeks 1-6 With Temozolomide & Radiation (N=2)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1: Selinexor 80mg on Weeks 1, 2, 4, 5 With Temozolomide & Radiation (N=3) | Dose Level 2: Selinexor 60mg Twice a Week on Weeks 1, 2, 4, 5 With Temozolomide & Radiation (N=6) | Dose Level 3: Selinexor 60mg Twice a Week, Weeks 1-6 With Temozolomide & Radiation (N=2)
Akathisia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (5) | 2 (3) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4) | 2 (2)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 3 (5) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Anxiety (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (3) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (3) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 3 (6) | 5 (6) | 1 (2)
Blurred vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Concentration impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Cushingoid (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 2 (3) | 0 (0)
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dysesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Dysphasia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Edema face (General disorders) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 1 (2) | 0 (0) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Fatigue (General disorders) | 3 (3) | 2 (3) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (8) | 5 (11) | 2 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 4 (8) | 2 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Infections and infestations - Other, COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (6) | 2 (3) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (9) | 6 (29) | 2 (5)
Lymphocyte count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (6) | 2 (6)
Platelet count decreased (Investigations) | 1 (2) | 4 (9) | 2 (7)
Seizure (Nervous system disorders) | 2 (4) | 3 (6) | 1 (2)
Serum amylase increased (Investigations) | 0 (0) | 1 (6) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Thrush (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vascular disorders - Other, DVT (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Weight gain (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 1 (4) | 3 (12) | 2 (11)
Wound complication (Injury, poisoning and procedural complications) | 1 (3) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-06-30): https://cdn.clinicaltrials.gov/large-docs/29/NCT04216329/Prot_SAP_002.pdf
  • Informed Consent Form (2023-02-22): https://cdn.clinicaltrials.gov/large-docs/29/NCT04216329/ICF_001.pdf